CLINICAL TRIAL: NCT04205708
Title: Screening Strategy for Early Diagnosis of Silicosis in At-Risk Populations in Oklahoma
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 10140
Record Dates: First submitted 2019-11-19; First posted 2019-12-19 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Silicosis; Pneumoconiosis; Silica
Keywords: silica; public health; early prevention; silicosis; screening; Oklahoma; lung disease; pulmonology; Pneumoconiosis; lung; dust exposure; occupational health; community health
MeSH Terms: conditions — Silicosis; Lung Diseases; Pneumoconiosis | interventions — Diagnostic Imaging; Respiratory Function Tests; Spirometry

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Tuberculosis test — Tuberculosis (TB) test: A blood sample is collected for lab testing to determine if you have tuberculosis (QuantiFeron test). Alternatively, the test is done by injecting a small amount of fluid (called tuberculin) into the skin on the lower part of the arm. A person given the tuberculin skin test must return within 48 to 72 hours to have a trained health care worker look for a reaction on the arm.
  Other Names: Mantoux skin test; QuantiFeron test
Diagnostic Test: Chest X-ray — Chest X ray: non-invasive medical test that helps physicians diagnose and treat medical conditions of the lungs and chest. The Chest X-ray will be done to check for abnormalities on the lungs. The test is non-invasive.
Diagnostic Test: Pulmonary Function Test — A pulmonary function test (PFT, spirometry) is a breathing test that measures how much air your lungs can hold as well as how hard and fast you can blow air out of your lungs. The test is not invasive and involves blowing into a machine.
  Other Names: Spirometry; Forced Spirometry

SUMMARY:
Silicosis, a preventable yet irreversible occupational lung disease, has an insidious onset with a latency period for diagnosis extending beyond 10 years from the initial exposure. The central hypothesis of this study is that silicosis cases may currently be going undetected. The long-term goal of this research is to determine the current prevalence and forecast the future prevalence of silicosis and other pneumoconiosis among working populations in Oklahoma and to assist the public health and the healthcare system in planning for a potential resurgence of silicosis.

ELIGIBILITY:
Inclusion Criteria:

* Male 30 years or older
* Past or present employment in dusty environment, exposed to dust at work
* Ability to consent and answer the questionnaire

Exclusion Criteria:

* Female
* Never exposed to dusty environment or never exposed to dust at work
* Inability to consent and answer the questionnaire
* Age 29 years or younger

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men Male gender identity
Study Population: Primary care clinic, community sample
  Participants will be recruited from waiting rooms or other common spaces at participating community health clinics.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Estimate of average cumulative respirable crystalline silica exposure (semi-quantitative) | Single point assessment at baseline survey
  Estimate of average cumulative respirable crystalline silica exposure (semi-quantitative)
Percentage of participants who report any exposure to silica | Single point assessment at baseline survey
  Percentage of participants who report any exposure to silica
Prevalence of silicosis among study group | Single point assessment at clinic visit
  Percentage of participants with confirmed diagnosis of silicosis

SECONDARY OUTCOMES:
Analysis to determine if any demographic, work history, or other trait correlates with increased silica exposure | Single point assessment at baseline survey
  Analysis to determine if any demographic, work history, or other trait correlates with increased silica exposure

CONTACTS AND LOCATIONS:
Overall Officials: Jad Kebbe, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers may request a deidentified dataset.
  The de-identified dataset may be shared between other investigators of the same institution as the PI, in accordance with University and Institutional Review Board policies.
  Any investigator not affiliated with the University of Oklahoma Health Sciences Center who desires access to a de-identified dataset may do so by coordinating a Data Use Agreement between the investigator's institution and the PI's institution.
  Datasets will only be released with an active Data Use Agreement or other similar agreement with the University of Oklahoma Health Sciences Center.
Time Frame: 2 years after publication
Access Criteria: Active Data Use Agreement or other similar agreement with the University of Oklahoma Health Sciences Center